CLINICAL TRIAL: NCT01204242
Title: IRB-HSR# 13957: IV Lidocaine for Patients Undergoing Primary Breast Cancer Surgery: Effects on Postoperative Recovery and Cancer Recurrence
Brief Title: IRB-HSR# 13957: IV Lidocaine for Patients Undergoing Primary Breast Cancer Surgery:
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Mohamed Tiouririne, MD, Associate Professor of Anesthesiology, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13957
Record Dates: First submitted 2010-09-15; First posted 2010-09-17 (Estimated); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): ALL subjects will receive lidocaine up to 1.5mg/kg IV (in the vein) as a rapid injection.
  Then the continuous IV infusion of the study medication (containing lidocaine 8 mg/ml or placebo) will be started and will continue for up to two hours in the recovery room.
  Interventions: Drug: Placebo
- Lidocaine (Experimental): ALL subjects will receive lidocaine up to 1.5mg/kg IV (in the vein) as a rapid injection.
  Then the continuous IV infusion of the study medication (containing lidocaine 8 mg/ml or placebo) will be started and will continue for up to two hours in the recovery room.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Placebo — ALL subjects will receive lidocaine up to 1.5mg/kg IV (in the vein) as a rapid injection.
  Then the continuous IV infusion of the study medication (containing lidocaine 8 mg/ml or placebo) will be started and will continue for up to two hours in the recovery room.
  Other Names: xylocaine
  Arms: Placebo
Drug: Lidocaine — ALL subjects will receive lidocaine up to 1.5mg/kg IV (in the vein) as a rapid injection.
  Then the continuous IV infusion of the study medication (containing lidocaine 8 mg/ml or placebo) will be started and will continue for up to two hours in the recovery room.
  Other Names: xylocaine
  Arms: Lidocaine

SUMMARY:
The purpose of this study is to determine whether a local anesthetic drug (lidocaine) given during anesthesia intravenously (IV) through a needle in your vein,), can:

1. Help decrease pain after surgery.
2. Have you need less pain medication.
3. Have less side effects like nausea and vomiting following your surgery.
4. Help to prevent chronic pain.
5. Affect recurrence of cancer after surgery.

DETAILED DESCRIPTION:
Pain after breast surgery is usually treated with narcotics; however, these are associated with a high incidence of side effects such as itching, nausea and vomiting, constipation, urinary retention and dizziness. Another modality for pain control is regional anesthesia; thoracic paravertebral blocks [TPVB] using local anesthetics are particularly appealing for breast surgery. They provide good pain control, possibly blunting surgical stress response, and decrease the need for anesthetic agent. However, TPVB are not widely used, and the inherent risk associated with their placement, such as pneumothorax, nerve injury, bleeding and infection, makes them less appealing to patients. From a pain management point of view, paravertebral blocks may be the optimal approach for reducing pain and opiate consumption after breast cancer surgery. In addition, retrospective data suggest a reduction in cancer recurrence if this technique is used. Unfortunately, this effective technique is not widely performed because of the risk of pneumothorax and is only used in some centers. Our intent is to study an alternative approach with fewer risks.

In this study, we will test the ability of intravenous lidocaine to provide pain relief after breast surgery. We base our hypothesis on a number of previous trials showing significant benefits of intravenous local anesthetics in the setting of abdominal surgery1-4.

Approximately 30 to 50% of patients will develop chronic pain following mastectomy5,6. It has been suggested that adequately treating pain in the immediate perioperative period will prevent chronic pain. Specifically, application of EMLA (local anesthetic) cream perioperatively during breast surgery has been shown to reduce the incidence of chronic pain development7. Perioperative administration of intravenous lidocaine may offer similar benefits. Therefore, we will study the incidence of chronic pain in our population after 6 months.

Finally, anesthetic choice during primary surgical intervention for cancer may affect recurrence and metastasis. A recent retrospective study suggests a profound reduction in recurrence in breast cancer patients receiving regional + general anesthesia as compared with general alone9. Similar data have been published in abstract form regarding recurrence after prostate surgery10. Also, Christopherson et al studied the long-term survival of 177 patients after resection of colon cancer in a trial of general anesthesia with and without epidural anesthesia and analgesia supplementation for resection of colon cancer. Epidural supplementation was associated with enhanced survival among patients without metastases before 1.46 years8. Although the mechanisms of this beneficial effect are unclear, attenuation of the surgical stress response, modulation of the inflammatory system, and/or decreased requirement for volatile anesthetics and opiates by regional anesthesia are possible mechanisms11. For example, the neural inputs activated during surgical stress may result in activation of promalignant pathways. Morphine has been shown to promote angiogenesis in a model of breast cancer, a key step in tumor development12. In addition, opiates interfere with natural killer cell function13. It is conceivable that the beneficial effect on recurrence might derive from low systemic level of local anesthetics attained during regional anesthesia. A number of studies have demonstrated significant reduction in opiate requirements and a decrease in the magnitude of stress response when local anesthetics are used intravenously1,3,4. If so, systemic administration would be a safer and a simpler way to reach the same goal. We therefore will compare the effect of local anesthetics given intravenously as compared with placebo on cancer recurrence rate.

ELIGIBILITY:
Inclusion Criteria:

1. informed consent
2. age older than 18 to 80 years (inclusive)
3. scheduled for mastectomy because of breast cancer
4. American Society of Anesthesiologists (ASA) physical classification classes I - III

Exclusion Criteria:

1. Allergy to local anesthetics, fentanyl or morphine
2. severe cardiovascular disease (myocardial infarction within 6 months), profoundly decreased left ventricular function (ejection fraction <40%) or high-grade arrhythmias
3. severe liver disease (known AST or ALT or billirubin >2.5 times the upper limit of normal)
4. renal impairment (creatinine clearance less than 60)
5. pregnant or breast feeding
6. patient is enrolled in another study or have been in one in the last 30 days

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2009-08-01 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2018-11-08 (Actual)

PRIMARY OUTCOMES:
opiate consumption | hospital discharge/ days 0-7
  We hypothesize that intraoperative use of intravenous lidocaine (as compared with placebo) will result in: decreased opiate consumption (primary endpoint), less pain, less fatigue and earlier postoperative discharge.

SECONDARY OUTCOMES:
chronic pain | 6 months after surgery
  We hypothesize that patients receiving IV lidocaine will report less pain than those in the placebo group at 6 months following surgery.
cancer recurrence | yearly for 5 years after surgery
  We hypothesize that patients in the IV lidocaine group will have a lower rate of cancer recurrence than those in the placebo group at 5 years following surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Tiouririne, MD, Principal Investigator — UVA Dept of Anesthesiology
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaba A, Laurent SR, Detroz BJ, Sessler DI, Durieux ME, Lamy ML, Joris JL. Intravenous lidocaine infusion facilitates acute rehabilitation after laparoscopic colectomy. Anesthesiology. 2007 Jan;106(1):11-8; discussion 5-6. doi: 10.1097/00000542-200701000-00007. PMID 17197840
- [Background] Herroeder S, Pecher S, Schonherr ME, Kaulitz G, Hahnenkamp K, Friess H, Bottiger BW, Bauer H, Dijkgraaf MG, Durieux ME, Hollmann MW. Systemic lidocaine shortens length of hospital stay after colorectal surgery: a double-blinded, randomized, placebo-controlled trial. Ann Surg. 2007 Aug;246(2):192-200. doi: 10.1097/SLA.0b013e31805dac11. PMID 17667496
- [Background] Groudine SB, Fisher HA, Kaufman RP Jr, Patel MK, Wilkins LJ, Mehta SA, Lumb PD. Intravenous lidocaine speeds the return of bowel function, decreases postoperative pain, and shortens hospital stay in patients undergoing radical retropubic prostatectomy. Anesth Analg. 1998 Feb;86(2):235-9. doi: 10.1097/00000539-199802000-00003. PMID 9459225
- [Background] Cassuto J, Wallin G, Hogstrom S, Faxen A, Rimback G. Inhibition of postoperative pain by continuous low-dose intravenous infusion of lidocaine. Anesth Analg. 1985 Oct;64(10):971-4. PMID 3898920
- [Background] Wallace MS, Wallace AM, Lee J, Dobke MK. Pain after breast surgery: a survey of 282 women. Pain. 1996 Aug;66(2-3):195-205. doi: 10.1016/0304-3959(96)03064-3. PMID 8880841
- [Background] Jung BF, Ahrendt GM, Oaklander AL, Dworkin RH. Neuropathic pain following breast cancer surgery: proposed classification and research update. Pain. 2003 Jul;104(1-2):1-13. doi: 10.1016/s0304-3959(03)00241-0. No abstract available. PMID 12855309
- [Background] Fassoulaki A, Sarantopoulos C, Melemeni A, Hogan Q. EMLA reduces acute and chronic pain after breast surgery for cancer. Reg Anesth Pain Med. 2000 Jul-Aug;25(4):350-5. doi: 10.1053/rapm.2000.7812. PMID 10925929
- [Background] Christopherson R, James KE, Tableman M, Marshall P, Johnson FE. Long-term survival after colon cancer surgery: a variation associated with choice of anesthesia. Anesth Analg. 2008 Jul;107(1):325-32. doi: 10.1213/ane.0b013e3181770f55. PMID 18635504
- [Background] Exadaktylos AK, Buggy DJ, Moriarty DC, Mascha E, Sessler DI. Can anesthetic technique for primary breast cancer surgery affect recurrence or metastasis? Anesthesiology. 2006 Oct;105(4):660-4. doi: 10.1097/00000542-200610000-00008. PMID 17006061
- [Background] Biki B MD, Sessler DI, Mascha E, Buggy DJ: Can Anaesthetic Technique for Radical Prostatectomy Surgery Affect Recurrence or Metastasis?, ASA Annual Meeting American Society of Anesthesiologists. San Francisco, 2007
- [Background] Ben-Eliyahu S, Page GG, Yirmiya R, Shakhar G. Evidence that stress and surgical interventions promote tumor development by suppressing natural killer cell activity. Int J Cancer. 1999 Mar 15;80(6):880-8. doi: 10.1002/(sici)1097-0215(19990315)80:63.0.co;2-y. PMID 10074922
- [Background] Farooqui M, Li Y, Rogers T, Poonawala T, Griffin RJ, Song CW, Gupta K. COX-2 inhibitor celecoxib prevents chronic morphine-induced promotion of angiogenesis, tumour growth, metastasis and mortality, without compromising analgesia. Br J Cancer. 2007 Dec 3;97(11):1523-31. doi: 10.1038/sj.bjc.6604057. Epub 2007 Oct 30. PMID 17971769
- [Background] Eisenstein TK, Hilburger ME. Opioid modulation of immune responses: effects on phagocyte and lymphoid cell populations. J Neuroimmunol. 1998 Mar 15;83(1-2):36-44. doi: 10.1016/s0165-5728(97)00219-1. PMID 9610671
- [Background] Apfel CC, Korttila K, Abdalla M, Kerger H, Turan A, Vedder I, Zernak C, Danner K, Jokela R, Pocock SJ, Trenkler S, Kredel M, Biedler A, Sessler DI, Roewer N; IMPACT Investigators. A factorial trial of six interventions for the prevention of postoperative nausea and vomiting. N Engl J Med. 2004 Jun 10;350(24):2441-51. doi: 10.1056/NEJMoa032196. PMID 15190136
- [Derived] Terkawi AS, Durieux ME, Gottschalk A, Brenin D, Tiouririne M. Effect of intravenous lidocaine on postoperative recovery of patients undergoing mastectomy: a double-blind, placebo-controlled randomized trial. Reg Anesth Pain Med. 2014 Nov-Dec;39(6):472-7. doi: 10.1097/AAP.0000000000000140. PMID 25275577